CLINICAL TRIAL: NCT03610880
Title: A Single Center, Randomized, Open-label, Two-arm, Parallel Design Study to Evaluate PK and Safety Profile of Multiple Ascending Oral Doses of Separately Using TG-2349 or DAG181 or TG-2349 Plus DAG181 in Healthy Chinese Volunteers
Brief Title: To Evaluate PK and Safety Profile of Oral MAD of Separately Using TG-2349, DAG181 or Combination in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongguan HEC TaiGen Biopharmaceuticals Co., Ltd. (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TGDAG-C-1
Record Dates: First submitted 2018-05-24; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Healthy Chinese Volunteers
Keywords: healthy Chinese volunteers; TG-2349; DAG181; pharmacokinetics; safety; multiple ascending oral doses
MeSH Terms: interventions — yimitasvir

STUDY DESIGN:
Intervention Model Description: randomized, open-label, two-arm, parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG-2349 (400 mg) plus DAG181 (200 mg) (Experimental): Dosing period 1 (Day 1 to 7): TG-2349 alone；Dosing period 2 (Day 8 to 14): TG-2349+DAG181
  Interventions: Drug: TG-2349 (400 mg) plus DAG181 (200 mg)
- DAG181 (200 mg) plus TG-2349 (400 mg) (Experimental): Dosing period 1 (Day 1 to 7): DAG181 alone；Dosing period 2 (Day 8 to 14): TG-2349+DAG181
  Interventions: Drug: DAG181 (200 mg) plus TG-2349 (400 mg)

INTERVENTIONS:
Drug: TG-2349 (400 mg) plus DAG181 (200 mg) — Dosing period 1 (Day 1 to 7): TG-2349 400 mg； Dosing period 2 (Day 8 to 14): TG-2349 400 mg + DAG181 200 mg
  Arms: TG-2349 (400 mg) plus DAG181 (200 mg)
Drug: DAG181 (200 mg) plus TG-2349 (400 mg) — Dosing period 1 (Day 1 to 7): DAG181 200 mg； Dosing period 2 (Day 8 to 14): TG-2349 400 mg + DAG181 200 mg
  Arms: DAG181 (200 mg) plus TG-2349 (400 mg)

SUMMARY:
To evaluate the drug-drug reactions between TG-2349 and DAG181, and the pharmacokinetics and tolerability profile in healthy Chinese volunteers to be the reference for protocol designs of subsequent clinical trials.

DETAILED DESCRIPTION:
This is a single center, randomized, open-label, two-arm, parallel design, phase I study that using TG-2349 or DAG181 alone, or TG-2349 plus DAG181 to evaluate the drug-drug reactions, the pharmacokinetics, and tolerability profile in healthy Chinese volunteers. The results will be the reference for protocol designs of subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Before starting the study, an informed consent form (ICF) approved by the Institute Review Board (IRB) is obtained from the subject or his/her legal representative；
2. Male or female, and 18 to 45 years of age inclusive when signing ICF；
3. Body mass index (BMI) in the range of 19.0 to 24.0 kg/m2 inclusive and male body weight ≥ 50 kg, female body weight ≥ 45 kg；
4. In general good physical and mental health status on basis of medical history review, physical examination and vital signs, 12-lead ECG, and laboratory results at screening；
5. For females, one of the following criteria must be fulfilled: (a) Had undergone surgical sterilization, or (b) Subjects of childbearing potential must satisfy the following criteria: Before group assignment, the urine pregnancy test is negative, and Subjects agree to use an approved contraceptive method (i.e. oral spermicidal agent, condoms, or intrauterine devices) during the entire study period (from Visit1 to Visit 2). Subject must also consent to keep the contraceptive method until 1 month after the study, and Breastfeeding is prohibited；
6. Male must be willing to use a reliable form of contraception (use of a condom or spouses using any of the above standards) during the entire study period (from Visit1 to Visit 2) and within 1 month after the study；
7. Have not used tobacco or nicotine-containing products within 1 month period to first dose of study drug；
8. Willing to abstain from caffeine- or xanthine-containing beverages, including coffee and tea, chocolate, alcohol, grapefruit juice, and Seville oranges juice before 24 hr and during the Stay-on Site period.

Exclusion Criteria:

1. Current, prior history, or family history of any disease of sudden cardiac death, myocardial ischemia, myocardial infarction, congestive heart failure, QT prolongation syndrome, hypokalemia, myocarditis, exertional dyspnea, cerebrovascular injury, venous thromboembolism；
2. Requires concomitant medication associated with increased QTc interval (i.e. Class I or III antiarrhythmic agents, refer to appendix 1) or with cardiac insufficiency；
3. Any abnormality on 12-lead ECG: PR>240 ms, PR<110 ms, QRS>110 ms, QTc>450 ms, or bradycardia ( heart rate < 50 beats/min) at screening or the day -1；
4. Any clinical significant abnormality on 12-lead ECG (i.e. atrioventricular block, TdT, other types of ventricular tachycardia, atrial fibrillation and ventricular flutter, clinical significant abnormality on T wave changes or any abnormality on 12-lead ECG that effects QTc intervals) at screening or the day -1；
5. Systolic pressure >140 mmHg or <90 mmHg, diastolic pressure >90 mmHg, pulse <50 beats/min or >100 beats/min at screening or the day -1；筛选或研究第-1天时收缩压>140 mmHg或<90 mmHg、舒张压>90 mmHg、脉搏<50次/分或>100次/分；
6. Any clinical significant abnormality on chest X-rays or abdominal ultrasound scan at screening (or within 2 weeks of signing the ICF)；
7. Positive serological test for hepatitis A (IgM anti-HAV), hepatitis B (HbsAg), hepatitis C (anti-HCV antibody), or syphilis at screening；
8. Pregnant or breastfeeding；
9. Any abnormal laboratory values (normal value ±10％) that are considered clinical significant by the Investigator at screening or the day -1；
10. Positive breath alcohol test or urine drug screen at screening or the day -1；
11. Current or prior history of any disease of diabetes, cardiovascular, hepatic or renal impairment；
12. Any dysphagia, malabsorption syndrome, or other gastrointestinal disturbances affecting drug absorption；
13. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy；
14. History of epileptic seizure, mental disorders affecting the subject's compliance with the protocol, suicidal risk, or a history of alcohol or illicit drug abuse；
15. Currently has any disease that seriously affects the immune system, for instance, human immunodeficiency virus (HIV) infection, hematological malignancy, solid cancer or splenectomy；
16. Allergy, hypersensitivity or allergic reaction to TG-2349 or its excipients, DAG181 or its excipients,or Sulfonamides；
17. History of surgery within 6 months prior to the first dose of study drug；
18. Received any hepatic enzyme inducers or hepatic enzyme inhibitors within 30 days prior to the first dose of study drug through medical history questionnaire (refer to appendix 2)；
19. Received any investigational drugs within 3 months prior to the first dose of study drug；
20. Received any prescription drugs, over-the-counter (OTC) drugs, or Chinese herbal medicines within 14 days prior to the first dose of study drug；
21. Received any nutritional supplies, including multivalent cations products (i.e. Ca-, Al-, Mg-, Fe-, and Zn-containing products, nutritional supplements, multi-vitamin, supplements for metals) within 7 days prior to the first dose of study drug；
22. History of alcohol misuse (14 units alcohol/ week: 1 unit equal to bear 285 mL, spirits 25 mL, or wine 100 mL)；
23. Blood donation ≥400 ml within 3 months prior to the first dose of study drug；
24. Any disease or situation that would affect the safety of study drug or pharmacokinetics profile by Investigators' judgments；
25. As determined by Investigator, a subject is not suitable to take part in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Cmax(ss) | 14 weeks
  Maximum Plasma Concentration in a stable state
Ctrough(ss) | 14 weeks
  Trough Plasma Concentration in a stable state
AUC(0-τ, ss) | 14 weeks
  Area Under the Plasma Concentration vs. Time Curve

SECONDARY OUTCOMES:
Cmax | 14 weeks
  Cmax: Maximum Plasma Concentration,
Ctrough | 14 weeks
  Ctrough: Trough Plasma Concentration
Tmax | 14 weeks
  Time at Which Maximum Plasma Concentration is Observed
AUC(0-24) | 14 weeks
  AUC(0-24): Area Under the Plasma Concentration vs. Time Curve 0-24 hours
Tmax(ss) | 14 weeks
  Tmax(ss): Time at Which Maximum Plasma Concentration is Observed in a stable state
λz | 14 weeks
  λz: Terminal disposition rate constant/terminal rate constant
AUC(0-last) | 14 weeks
  AUC(0-last): Area Under the Plasma Concentration vs. Time Curve 0 - the last dose
AUC(0-inf) | 14 weeks
  AUC(0-inf): Area Under the Plasma Concentration vs. Time Curve 0 - infinity
MRT | 14 weeks
  MRT: mean residence time
CL/F | 14 weeks
  CL/F: total clearance rate
V/F | 14 weeks
  V/F: apparent volume of distribution
DF | 14 weeks
  DF=(Cmax - Ctrough) / (AUCss /τ)
12-lead ECG | 19 weeks
  including heart rate, RR, PR, QRS, QT, QTc；
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 19 weeks
  CTCAE v4.0
blood pressure (mmHg) | 19 weeks
  Vital signs
pulse (beats/ min) | 19 weeks
  Vital signs
respiratory rate (breaths/ min) | 19 weeks
  Vital signs
body temperature (oC) | 19 weeks
  Vital signs
General Appearance Physical examination | 19 weeks
  Physical examination
Skin Physical examination | 19 weeks
  Physical examination
Head and Neck Physical examination | 19 weeks
  Physical examination
Chest region Physical examination | 19 weeks
  Physical examination
Abdominal region Physical examination | 19 weeks
  Physical examination
Back region Physical examination | 19 weeks
  Physical examination
Extremities Physical examination | 19 weeks
  Physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Xu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China